CLINICAL TRIAL: NCT03871751
Title: Evaluating the Effectiveness of Home-based SSP on Individuals With PWS
Brief Title: Home-based SSP on Individuals With PWS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources to complete study as planned
Sponsor: Indiana University (Other)
Collaborators: Integrated Listening Systems (Unknown)
Responsible Party: Principal Investigator, Jacek Kolacz, Assistant Research Scientist, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1807300643
Record Dates: First submitted 2019-02-25; First posted 2019-03-12 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Prader-Willi Syndrome
Keywords: Polyvagal Theory; Social Behavior; Hyperacusis; Prosody; Auditory intervention
MeSH Terms: conditions — Prader-Willi Syndrome; Social Behavior; Hyperacusis

STUDY DESIGN:
Intervention Model Description: All participants will receive the auditory intervention.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safe and Sound Protocol (Experimental): All child participants will participate in 1 pre-intervention assessment and 1 post-intervention assessment. The auditory intervention (i.e., Safe and Sound Protocol, SSP) will last for 1 hour per day, for 5 consecutive days.
  Interventions: Behavioral: Safe and Sound Protocol

INTERVENTIONS:
Behavioral: Safe and Sound Protocol — The auditory intervention will consist of listening to computer-altered acoustic stimulation, designed to modulate the frequency band of vocal music passed to the participant. The frequency characteristics of the acoustic stimulation are selected to emphasize the relative importance of specific frequencies in conveying the information embedded in human speech. Modulation of the acoustic energy within the frequencies of human voice, similar to an exaggerated vocal prosody, are hypothesized to recruit and modulate the neural regulation of the middle ear muscles and to functionally reduce sound hypersensitivities and improve auditory processing.
  Other Names: Listening Project Protocol

SUMMARY:
The Polyvagal Theory focuses on how function and structure changed in the vertebrate autonomic nervous system during evolution. The theory is named for the vagus, a major cranial nerve that regulates bodily state. As a function of evolution, humans and other mammals have a "new" vagal pathway that links the regulation of bodily state to the control of the muscles of the face and head including the middle ear muscles. These pathways regulating body state, facial gesture, listening (i.e., middle ear muscles), and vocal communication collectively function as a Social Engagement System (SES). Because the Social Engagement System is an integrated system, interventions influencing one component of this system (e.g., middle ear muscles) may impact on the other components.

Individuals with Prader-Willi Syndrome (PWS) exhibit many behaviors that are consistent with a compromised Social Engagement System. Atypical function of the Social Engagement System results in problems associated with state regulation (e.g., impulsivity, tantrums, and difficulty with change in routine), ingestion (e.g., difficulties in sucking at birth, hyperphagia), coordination of suck/swallow/breathe, intonation of vocalizations, auditory processing and hypersensitivity, and socialization. The investigatiors propose to confirm that several features of the behavioral phenotype of PWS may be explained within the context of a dysfunctional SES, which may be partially rehabilitated via an intervention designed as a 'neural exercise' of the SES (i.e., the Safe and Sound Protocol, "SSP").

Specific Aims:

Aim I: To demonstrate the effectiveness of the Safe and Sound Protocol (SSP) on improvement of social and regulation behaviors in individuals with PWS.

Aim II: To evaluate a new methodology for collecting and evaluating vocal samples for analyses of prosody, one of the indices of the functioning of the SES.

ELIGIBILITY:
Inclusion Criteria:

1. Child participants must meet criteria for Prader-Willi Syndrome (per parent membership in Prader-Willi Parent Support Group).
2. Child participants must be between ages 3-17 years. Parent must be 18 years or older.
3. Child participants must have normal hearing (confirmed via parental report on Qualtrics questionnaire)

Exclusion Criteria:

1) Child participants who are hearing-impaired (without correction)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sensory sensitivities at 1 week | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention)
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)

SECONDARY OUTCOMES:
Change from baseline in disruptive behavior at 1 week | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention)
  Developmental Behavior Checklist (DBC2) (questionnaire)
Change from baseline in social behavior at 1 week | post-intervention (within 1 week after intervention)
  Safe and Sound Protocol (SSP) Parent Questionnaire
Change from baseline in Foundational Abilities (balance, gross & fine motor control, sensory, social/emotional, auditory/language and attention/organization and sleep) at 1 week | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention)
  Measure of Foundational Abilities (MFA) questionnaire
Change from baseline in prosody at 1 week | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention)
  Prosody assessment of recorded speech

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kolacz, PhD, Principal Investigator — Indiana University/Kinsey Institute
Locations (1):
- Integrated Listening Systems, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porges SW. The polyvagal theory: phylogenetic substrates of a social nervous system. Int J Psychophysiol. 2001 Oct;42(2):123-46. doi: 10.1016/s0167-8760(01)00162-3. PMID 11587772
- [Background] Porges SW, Bazhenova OV, Bal E, Carlson N, Sorokin Y, Heilman KJ, Cook EH, Lewis GF. Reducing auditory hypersensitivities in autistic spectrum disorder: preliminary findings evaluating the listening project protocol. Front Pediatr. 2014 Aug 1;2:80. doi: 10.3389/fped.2014.00080. eCollection 2014. PMID 25136545